CLINICAL TRIAL: NCT07098234
Title: Determination of the Effect of Vitamin-D as an Adjuvant to Phototherapy in Reduction of Indirect Serum Bilirubin Among Neonates With Exaggerated Physiological Hyperbilirubinemia.
Brief Title: Effect of Vitamin-D as an Adjuvant to Phototherapy in Reduction of Indirect Serum Bilirubin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dr-Hafsah-LHR
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Hyperbilirubinemia
MeSH Terms: conditions — Hyperbilirubinemia | interventions — Cholecalciferol; Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D3 group (Experimental): Neonates were given vitamin D3 (cholecalciferol) in an oral drops formulation (400 IU/drop), at a dose of 400 IU once a day for 72 hours as an adjuvant therapy to phototherapy.
  Interventions: Drug: Vitamin D3; Procedure: Phototherapy
- Phototherapy group (Experimental): Neonates received only phototherapy for 72 hours.
  Interventions: Procedure: Phototherapy

INTERVENTIONS:
Drug: Vitamin D3 — Neonates were given vitamin D3 (cholecalciferol) in an oral drops formulation (400 IU/drop), at a dose of 400 IU once a day until the serum bilirubin level was out of phototherapy range or a maximum of 72 hours as an adjuvant therapy to phototherapy.
  Arms: Vitamin D3 group
Procedure: Phototherapy — Neonates received only phototherapy until the serum bilirubin level was out of phototherapy range or a maximum of 72 hours.

SUMMARY:
The study aimed at filling the gaps by evaluating the effectiveness of vitamin-D as an adjuvant to phototherapy in reduction of indirect serum bilirubin among neonates with exaggerated physiological hyperbilirubinemia.

DETAILED DESCRIPTION:
If vitamin-D has been found effective as an adjuvant to phototherapy in the treatment of exaggerated physiological hyperbilirubinemia, it may help to reduce the serum bilirubin level rapidly. It may also reduce the complications by shortening the duration of phototherapy to offer better patient compliance and better patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Newborns of any gender
* Age of 3rd day of life to 8th day of life
* Gestation age ≥37 to ≤42 weeks
* Total serum bilirubin level more than 12.9 mg/dL
* Weight > 2.5 kg

Exclusion Criteria:

* Congenital defects (on physical examination)
* Large for gestational age infant
* Rh Incompatibility (were excluded on basis of blood grouping of mother and baby)
* ABO Incompatibility (were excluded on basis of blood grouping of mother and baby)
* Neonatal sepsis

Ages: 3 Days to 8 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Bilirubin reduction comparison | 72 hours
  Net reductions in bilirubin levels in two groups after 72 hours were compared.

CONTACTS AND LOCATIONS:
Overall Officials: Hafsah Naz, Principal Investigator — Mayo Hospital, Lahore, Pakistan; Muhammad Ashfaq, Principal Investigator — Mayo Hospital, Lahore, Pakistan
Locations (1):
- Mayo Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
The data can be shared on a reasonable request.